CLINICAL TRIAL: NCT06815237
Title: Acute Effects of Ketone Supplementation and Alcohol on Brain Metabolism
Brief Title: Effects Ketone Supplement and Alcohol on Brain Metabolism
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 857606; R21AA031088-01A1 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ketosis; Alcohol Drinking; MRI
Keywords: ketone supplement
MeSH Terms: conditions — Ketosis; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will randomly receive each intervention once: ketone supplement, alcohol beverage, and no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketone Supplement (Experimental): Subjects will receive ketone supplement once by mouth, 20g of kentones.
  Interventions: Dietary Supplement: Kenetik
- Alcohol beverage (Experimental): Alcohol lab, participants will receive ethanol drinks that are dose-adjusted for body weight and sex differences in pharmacokinetics and calculated to obtain a final breath alcohol concentration of 0.050%
  Interventions: Other: Alcohol beverage
- No Intervention (No Intervention): No intervention will be given

INTERVENTIONS:
Dietary Supplement: Kenetik — Ketone supplement is randomly given once.
  Other Names: D-Beta-hydroxybutyric acid and R-1,3 butanediol; Ketone supplement
  Arms: Ketone Supplement
Other: Alcohol beverage — Alcohol beverage is randomly given once. Participants will receive the alcohol beverage that dose-adjusts for body weight and sex differences in pharmacokinetics and calculated to obtain a final breath alcohol concentration of 0.050%
  Other Names: Ethanol
  Arms: Alcohol beverage

SUMMARY:
The research study is being conducted to better understand the effects of ketones and alcohol on brain functioning and brain metabolism. Participants will be asked to undergo three identical MRI visits after three single-dose interventions: (1) drink a ketone supplement drink, (2) drink an alcoholic beverage, (3) no intervention. These interventions will be randomly assigned (meaning everyone receives all 3 interventions, but in different orders).

DETAILED DESCRIPTION:
Screening Visit: Participants will complete a screening visit at the CSA (Center for Studies of Addiction). At the visit participants will be asked to show legal photo identification and undergo a breath alcohol test to ensure a breath alcohol concentration (BrAC) of <0.000%, to ensure that the participant is not intoxicated, which would make it difficult to provide informed consent. Participants will be given the informed consent form to read, which a study staff member will then review, as well as provide an explanation of the study protocol, risks, potential benefits, and alternative treatments. Following resolution of any questions, participants will be asked to sign the consent form and an entire copy of it will be given to the participants. The participant will be reminded that signing the consent form represents their willingness to participate in the study but that the subsequent screening process will determine their eligibility to do so.

Next, the participant will meet with a study clinician who will obtain a medical history and conduct a physical examination. Trained staff will measure subjects' weight, height, and vital signs (blood pressure and heart rate). Study staff trained in phlebotomy will draw approximately 3 tablespoons (44 mL) of blood for baseline laboratory measure. Baseline laboratory samples will include:

* Complete blood count (CBC)
* Blood chemistries (i.e., standard blood work and lipids)
* Urinalysis
* Urine toxicology (presence of psychoactive drugs)
* Urine pregnancy test for women In cases where blood samples are drawn and potential lab errors or abnormal findings occur, subjects will be asked to provide an additional blood sample to repeat the test(s).

Study staff will complete the following assessments with participants during Consent/Screening:

* Sociodemographic/general participant information: An assessment of medical history, personal and family history of alcohol use disorder, marital status, educational and occupational information, and substance abuse treatment history will be obtained, along with the individual's self-identified ancestry.
* A structured diagnostic psychiatric interview for DSM-5, which will be used to identify current substance use- and psychiatric disorders.
* Timeline Follow-Back (TLFB) is a 90-day assessment of use of alcohol, opioids, caffeine, nicotine, marijuana, cocaine, amphetamine, methamphetamine, and benzodiazepines.
* MRI safety form: This standard assessment form, created by the Department of Radiology at the Hospital of the University of Pennsylvania, assesses the history of specific prostheses, surgical implants, and other MRI contraindications.
* Oral HIV test: participants will be administered an oral HIV test. If the HIV test positive, study staff will inform the participants of the results, counsel the participants regarding the need to confirm the finding with a blood test and to avoid potential exposure of others to HIV, and draw an additional 1/2 tablespoon of blood to conduct a confirmatory HIV blood test. If the blood test is positive for HIV, the participants will be referred for medical care and given a copy of the test to provide to the doctor for the follow-up visit.

After the screening visit is complete, staff will call participants within 5 business days to let them know whether or not the study is a good fit. If it is a good fit for staff will schedule the 3 study lab visits.

Study lab visits: Staff will contact the participant the day before the lab visit to take the breakfast order, snack order, and tell subjects if they need to take a Lyft into the study visit located at Stellar Chance Laboratories (440 Curie Blvd.). On the lab visit that participants receive alcohol beverages, they will need to take a Lyft to the visit and back home after the visit.

Each visit will start at approximately 8:30 am, and participants will meet staff at Stellar chance Lab. They will be asked to not eat or drink anything except water after midnight the day before and on the day of each of the study lab visits. Staff will provide a light breakfast,

Table 2. Timeline of events on Lab days Approximate time Study procedure 08:30 AM Participant arrives at the study site and breathalyzer (BrAC must be 0.000) 8:35 AM Vital signs, finger stick for blood glucose, and ketone levels 8:40 AM Urine sample for UDS and urine pregnancy test if you are a woman who is able to become pregnant. 8:45 AM Light breakfast 9:00 AM Staff will review with you any recently used drugs, alcohol, medications, or vitamins since your last visit. 9:45 AM Administration of KS (20g), or alcohol, or no intervention 10:00AM MRI 11:30 AM Breathalyzer, finger stick for blood glucose, and ketone levels 11:45 AM Snack 12:20 AM Breathalyzer (repeated until below 0.020), finger stick for blood glucose (repeated if glucose is below 70 mg/dl, until it returns to normal). 12:30 AM Once BrACH is below 0.020 and blood glucose levels return to normal levels a study clinician will meet with you to ask you some questions and complete a brief sobriety assessment to make sure it is safe for you to go home.

Follow-up (~5 minutes): On the first business day following the study visits, participants will receive a follow-up phone call from study staff to ask about any changes to their health and to ensure that they did not experience any side effects from the MRI scan or other laboratory procedures. If the next business day falls on a holiday, then the follow-up call may occur on the next business day.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and commit to completing study procedures.
2. Reported on at least one day in the month before consent of consuming 2 or more standard alcoholic drinks on a single day.

Exclusion Criteria:

1. Unwilling or unable to refrain from the use of psychoactive medications, medication that may affect study results, and or alcohol, within 24 hours of the Alcohol lab, and MRI procedures (self-report, medical history, UDS, and breathalyzer).
2. Current DSM-5 diagnosis of a major psychiatric disorder (other than marijuana and nicotine use disorders) as identified by clinical examination or structured interview that could interfere with study participation or make it hazardous for the subject.
3. Currently taking a medication that could interfere with study participation or make it hazardous for the subject to participate. (e.g., anticholinergics; antipsychotics; psychotropic drugs not otherwise specified)
4. Positive urine drug screen positive for all substances but marijuana on study visits (may be repeated once and if the result is negative on repeat it is not exclusionary).
5. A current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation that could interfere with study participation or make it hazardous for the subject to do so (e.g., bleeding disorder, pancreatitis, epilepsy, liver disease, kidney disease, or diabetes as determined by history and clinical exam); ALAT or ASAT concentration greater than 3 times the upper limit of normal (ULN), or bilirubin above the ULN. (Note-abnormal laboratory tests during screening may be repeated once).
6. Current, major gastrointestinal (GI) diseases, such as: GERD, Crohn's disease, Irritable bowel syndrome, Ulcerative colitis, Celiac disease Diverticulitis, or other clinically significant physical disease that may interfere with the intake of the Ketone Supplement based on medical history, and evaluation of the Study Physician.
7. Head trauma with loss of consciousness for more than 30 minutes (self-report, medical history).
8. Pregnant or breast-feeding
9. Weight greater than 250lbs (Need to cap amount of alcohol give based on weight to individuals).
10. Self-reported claustrophobia
11. Contraindications to MRI (e.g., metal in the body that cannot be removed and is not MRI compatible).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
To examine the acute effects of ketone supplements compared to no intervention on Nicotinamide adenine dinucleotide levels in the brain. | 60 minutes
  Use MRI imaging to measure the amount of Nicotinamide adenine dinucleotide levels in the brain measured in mmol/L in participants after receiving ketone supplement intervention compared to no intervention.
To examine the acute effects of ketone supplements compared to no intervention on brain Glutamate levels. | 45 minutes
  Use MRI imaging to measure the amount of Glutamate levels in the brain measured in mmol/L in participants after receiving ketone supplement intervention compared to no intervention.
To examine the acute effects of ketone supplements compared to no intervention on brain Gamma-aminobutyric acid levels. | 75 minutes
  Use MRI imaging to measure the amount of Gamma-aminobutyric acid levels in the brain measured in mmol/L in participants after receiving ketone supplement intervention compared to no intervention.

SECONDARY OUTCOMES:
To examine the acute effects of alcohol (dose adjusted by weight) compared to no intervention on Nicotinamide adenine dinucleotide levels in the brain. | 60 minutes
  Use MRI imaging to measure the amount of Nicotinamide adenine dinucleotide levels in the brain measured in mmol/L in participants after receiving an alcohol (dose adjusted by weight) intervention compared to no intervention.
To examine the acute effects of alcohol (dose adjusted by weight) compared to no intervention on brain Glutamate levels. | 45 minutes
  Use MRI imaging to measure the amount of Glutamate levels in the brain measured in mmol/L in participants after receiving an alcohol (dose adjusted by weight) intervention compared to no intervention.
To examine the acute effects of alcohol (dose adjusted by weight) compared to no intervention on brain Gamma-aminobutyric acid levels. | 75 minutes
  Use MRI imaging to measure the amount of Gamma-aminobutyric acid levels in the brain measured in mmol/L in participants after receiving an alcohol (dose adjusted by weight) intervention compared to no intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde Wiers, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Studies of Addiction, Philadelphia, Pennsylvania, United States